CLINICAL TRIAL: NCT03771157
Title: Serologic Response to a New Recombinant, Adjuvanted Herpes Zoster Vaccine in Patients With Chronic Lymphocytic Leukemia and Waldenström Macroglobulinemia Treated With First-Line BTK Inhibitors - A Pilot Study
Brief Title: Serologic Response to SHINGRIX Vaccine in Patients With CLL and WM Treated With BTK Inhibitors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jonathan Friedberg, Director of the Wilmot Cancer Institute, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003112
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Waldenstrom Macroglobulinemia (WM)
Keywords: shingles vaccine (Shingrix); Chronic lymphocytic leukemia (CLL); Waldenstrom macroglobulinemia (WM); Pilot Study
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shingrix shingles vaccine treatment (Experimental): On day one, patients will receive the first of two doses of the Shingrix vaccine administered as an injection into the muscle in their upper arm. The second dose of vaccine will be administered as an injection to their upper arm approximately 2 months after the first dose.
  Interventions: Drug: Shingrix vaccine

INTERVENTIONS:
Drug: Shingrix vaccine — On day one, patients will receive the first of two doses of the Shingrix vaccine administered as an injection into the muscle in their upper arm. The second dose of vaccine will be administered as an injection to their upper arm approximately 2 months after the first dose.
  Other Names: Herpes Zoster Vaccine Recombinant, Adjuvanted

SUMMARY:
The primary objective of the study is to assess the capability of a patient with Chronic Lymphocytic Leukemia (CLL) or Waldenström Macroglobulinemia (WM) to generate an immune response to the Shingrix vaccine under first-line BTK inhibitors.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and Waldenstrom's macroglobulinemia (WM) are known risk factors for zoster reactivation, commonly called shingles. Although a recently FDA-approved recombinant, adjuvanted herpes zoster vaccine (Shingrix) is currently being offered to these populations, no study has specifically evaluated them.

The purpose of the study is to complete a single-arm trial evaluating if patients with CLL or WM, while on treatment with first-line BTK inhibitors, can achieve immunologic response to Shingrix. If effective, this will result in a new, well-tolerated shingles prevention strategy for these patients.

The primary objective is to assess the capability to mount a humoral immune response to Shingrix in patients with CLL or WM under first-line BTK inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* They are at least 50 years of age;
* Have been diagnosed with chronic lymphocytic leukemia (CLL) OR Waldenström's macroglobulinemia (WM)
* Have been on first-line BTK inhibitor (ie ibrutinib or acalabrutinib) for at least 3 months,
* Prior treatment with single agent rituximab is permitted if last dose was administered over one year ago;
* Have at least a one-year life expectancy;
* Have a history of varicella (chicken-pox) OR lived in the US or any endemic country for > 30 years.
* Prior radiation therapy is allowed

Exclusion Criteria:

* They have a known hypersensitivity to a vaccine component;
* Had herpes zoster reactivation within the past year;
* Had received or were scheduled to receive a live virus vaccine in the period from 4 weeks prior to Dose 1 through 28 days post-second dose;
* Had received or were scheduled to receive an inactivated vaccine in the period ranging from 7 days prior to Dose 1 through 7 days post- second dose;
* Are unable to give informed consent;
* Have absolute lymphocyte counts greater than 20,000 X 109/L;
* Are receiving treatment for CLL or WM with an additional agent other than a BTK inhibitor;
* Had rituximab treatment within a year prior to study start;
* Had prior chemotherapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Friedberg, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shingrix Vaccine
Started | 32 (33 subjects consented, 1 subject withdrew before completing study procedures leaving 32 Started Subjects)
Completed | 31
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Shingrix Vaccine: On day one, patients will receive the first of two doses of the Shingrix vaccine administered as an injection into the muscle in their upper arm. The second dose of vaccine will be administered as an injection to their upper arm approximately 2 months after the first dose. Antibody and cellular response to vaccination will be assessed at 4 weeks and 24 months after the second dose.
Arm/Group | Shingrix Vaccine
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  50 to 65 years | 12
  > 65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Humoral Response to Vaccination 4 Weeks After the Second Vaccine Administration
Description: Vaccine response, as determined by blood antibody levels to the varicella virus glycoprotein E subunit (anti-gE); Baseline is defined as pre-vaccination anti-gE titer in seropositive subjects, and the lower limit of detection in seronegative subjects
Time Frame: 4 weeks following the second vaccination, at approximately 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Shingrix Vaccine: On day one, patients will receive the first of two doses of the Shingrix vaccine administered as an injection into the muscle in their upper arm. The second dose of vaccine will be administered as an injection to their upper arm approximately 2 months after the first dose. Antibody and cellular response to vaccination will be assessed at 4 weeks after the second dose.
Arm/Group | Shingrix Vaccine
Number analyzed (Participants) | 32
Participants | 24

2. Secondary Outcome: Number of Participants With Cellular Response to Vaccination 4 Weeks After the Second Vaccine Administration
Description: Cellular response, as determined by measuring VZgE-specific T-cell responses in blood, 4 weeks after the second vaccine administration.
Time Frame: 4 weeks following the second vaccination, at approximately 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shingrix Vaccine
Number analyzed (Participants) | 32
Participants | 26

3. Other Pre Specified Outcome: Number of Participants With Humoral Response to Vaccination 2 Years After the Second Vaccine Administration
Description: as for outcome 1
Time Frame: 2 years following second vaccination, approximately 26 months from day 1
Measure: Count of Participants; unit: Participants
Groups:
- Shingrix Vaccine: On day one, patients will receive the first of two doses of the Shingrix vaccine administered as an injection into the muscle in their upper arm. The second dose of vaccine will be administered as an injection to their upper arm approximately 2 months after the first dose. Antibody and cellular response to vaccination will be assessed at 24 months after the second dose.
Arm/Group | Shingrix Vaccine
Number analyzed (Participants) | 31
Participants | 13

4. Other Pre Specified Outcome: Number of Participants With Cellular Response to Vaccination 2 Years After the Second Vaccine Administration
Description: Cellular response, as determined by measuring VZgE-specific T-cell responses in blood, 2 years after the second vaccine administration.
Time Frame: 2 years following second vaccination, approximately 26 months from day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Shingrix Vaccine
Number analyzed (Participants) | 31
Participants | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day one to four weeks after the second vaccine administration, up to approximately 3 months.
Description: Only adverse events grade 3 and greater will be collected. Adverse events were obtained through medical chart review and self-reporting by participants.
Arm/Group | Shingrix Vaccine
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shingrix Vaccine (N=32)
Atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03771157/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03771157/ICF_000.pdf